CLINICAL TRIAL: NCT02308839
Title: Study of the GORE® EXCLUDER® Endoprosthesis in the Treatment of Infra-renal Abdominal Aortic Aneurysms
Brief Title: GORE® EXCLUDER® Endoprosthesis French Mandatory Registry
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: FPR12-02
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aneurysm; Aorta; Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GORE® EXCLUDER® Endoprosthesis — Endovascular therapy to treat abdominal aortic aneurysms

SUMMARY:
This is a French Registry mandated by the French National Health Authority assessing long-term (5-years) safety of the GORE® Excluder® Endoprosthesis in the treatment of infra-renal Abdominal Aortic Aneurysms (AAA).

DETAILED DESCRIPTION:
The use of abdominal aortic endoprostheses makes the treatment of infra-renal abdominal aortic aneurysms possible, with implantation via the femoral artery, thus avoiding a very invasive surgical procedure. The French National Authority for Health requires a 5-year follow-up as part of the renewal for reimbursement for these endoprostheses.

ELIGIBILITY:
Inclusion Criteria:

* Any patients requiring abdominal aortic stenting for the treatment of an unruptured infra-renal aortic abdominal aneurysm.

Exclusion Criteria:

* Patients whose clinical follow-up is not possible, i.eg, patient who cannot return for control visits (e.g. patients living abroad).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring treatemtn with an endoprosthesis for the treatment of an unruptured infra-renal aortic abdominal aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Steinmetz, Prof, Principal Investigator — Centre Hospitalier Universitaire du Bocage
Locations (1):
- Centre Hospitalier de Dijon, Dijon, France

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE® EXCLUDER® AAA Endoprosthesis: GORE® EXCLUDER® AAA Endoprosthesis
Period: Overall Study
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Started | 181
Completed | 72
Not Completed | 109

BASELINE CHARACTERISTICS:
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 162
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Survived at 5 Years
Description: Kaplan-Meier estimate of participant survival at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage of participants alive
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Percentage of participants alive | 76

2. Secondary Outcome: Percentage of Participants Free From Endoleak at 5 Years
Description: Kaplan-Meier estimate of participant freedom from endoleak (Type I, II and III) at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage free from endoleak
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Percentage free from endoleak | 72

3. Secondary Outcome: Percentage of Participants Free From Migration at 5 Years
Description: Kaplan-Meier estimate of participant freedom from migration at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage free from migration
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 178
Percentage free from migration | 100

4. Secondary Outcome: Percentage of Participants Free From Aneurysm Diameter Growth at 5 Years
Description: Kaplan-Meier estimate of participant freedom from aneurysm diameter growth at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage free from aneurysm growth
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 156
Percentage free from aneurysm growth | 77

5. Secondary Outcome: Percentage of Participants Free From Aneurysm Related Mortality at 5 Years
Description: Kaplan-Meier estimate of participant freedom from aneurysm related mortality at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage free from mortality
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Percentage free from mortality | 99

6. Secondary Outcome: Percentage of Participants Free From Endovascular or Surgical Re-intervention at 5 Years
Description: Kaplan-Meier estimate of participant freedom from endovascular or surgical re-intervention at 5 years
Time Frame: 5 years
Measure: Number; unit: Percentage free from re-intervention
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Percentage free from re-intervention | 75

7. Secondary Outcome: Percentage of Participants Free From Surgical Conversion at Procedure
Description: Participant freedom from surgical conversion at procedure
Time Frame: Index Procedure
Measure: Number; unit: Percentage free from conversion
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
Number analyzed (Participants) | 181
Percentage free from conversion | 100

ADVERSE EVENTS:
Time Frame: Five year follow-up
Groups:
- GORE® EXCLUDER® AAA Endoprosthesis: GORE® EXCLUDER® AAA Endoprosthesis Registry conducted for reimbursement in France, and no MedDRA coding was required.
Arm/Group | GORE® EXCLUDER® AAA Endoprosthesis
All-Cause Mortality (participants affected / at risk) | 35/181
Serious Adverse Events (participants affected / at risk) | 69/181
Other Adverse Events (participants affected / at risk) | 89/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® EXCLUDER® AAA Endoprosthesis (N=181)
Device Related (General disorders) | 6
Procedure Related (General disorders) | 10 — Procedure Related but not Device Related
Aneurysm Related (General disorders) | 17 — Aneurysm Related but not Device Related or Procedure Related
Other (General disorders) | 46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® EXCLUDER® AAA Endoprosthesis (N=181)
Device Related (General disorders) | 5
Procedure Related (General disorders) | 17 — Procedure Related but not Device Related
Aneurysm Related (General disorders) | 63 — Aneurysm Related but not Device Related or Procedure Related
Other (General disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-02-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02308839/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT02308839/SAP_001.pdf